CLINICAL TRIAL: NCT01435538
Title: The Impact of Care Pathways on Interprofessional Teamwork: an International Cluster Randomized Controlled Trial
Brief Title: European Quality of Care Pathways Study on the Effect of Care Pathways on Interprofessional Teamwork (EQCP-TEAM)
Acronym: EQCP-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kris Vanhaecht (Other)
Collaborators: KU Leuven (Other); University of Eastern Piedmont (Other)
Responsible Party: Sponsor-Investigator, Dr. Kris Vanhaecht, Secretary General, European Pathway Association
Organization: European Pathway Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPA-EQCP-003
Record Dates: First submitted 2011-09-15; First posted 2011-09-16 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Proximal Femur Fracture
Keywords: interprofessional teamwork; care pathways; team communication; team coordination; Chronic Obstructive Pulmonary Disease Teams; Proximal Femur Fracture Teams
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Proximal Femoral Fractures | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care pathway teams. (Experimental): In this experimental arm, the interprofessional teams will develop and implement a care pathways.
  Interventions: Behavioral: Care pathway.
- Usual care teams. (No Intervention): In the no intervention arm, the interprofessional teams will deliver usual care without implementing the intervention.

INTERVENTIONS:
Behavioral: Care pathway. — The intervention group will implement a care pathway for PFF or COPD containing three active components: a formative evaluation of the actual teams' performance, a set of evidence based key interventions and a training in pathway-development.
  Arms: Care pathway teams.

SUMMARY:
Care pathways are complex interventions to support the interprofessional team in the redesign of their care process. This international cluster randomised trial will analyse the impact of the development and implementation of care pathways on the interprofessional teamwork.

DETAILED DESCRIPTION:
Background Although care pathways are often said to promote teamwork, high-level evidence that supports this statement is lacking. The objective of the European Quality of Care Pathway (EQCP) study is therefore to study the impact of care pathways on interprofessional teamwork.

Methods/design An international post-test-only cluster Randomized Controlled Trial (cRCT), combined with process evaluations, will be performed in Belgium, Ireland, Italy and Portugal. Teams caring for Proximale Femur Fracture (PFF) patients and patients hospitalized with an exacerbation of Chronic Obstructive Pulmonary Disease (COPD) will be randomized into an intervention and control group. The intervention group will implement a care pathway for PFF or COPD containing three active components: a formative evaluation of the actual teams' performance, a set of evidence based key interventions and a training in pathway-development. The control group will provide usual care. As effect measures a set of team input, process and output indicators will be used. Main outcome indicator is the team process indicator relational coordination. Next to these, process measures will be used to evaluate the implementation process. In total, 132 teams agreed to participate, of which 68 were randomly assigned to the intervention group and 64 to the control group. Based on power analysis, a sample of 475 team members per arm is required. To analyze results, multilevel analysis will be performed.

Discussion The EQCP-study on teamwork is the first cluster-randomized controlled trial on the impact of care pathways on interprofessional teamwork. Results from our study will enhance understanding on the active components of care pathways. Through this, preferred implementation strategies can be defined.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion on cluster level requires the written agreement to participate form the hospital management, the medical head of the division and the head nurse
* Next to this, they have to agree that they will not develop and implement a care pathway for COPD- exacerbation of PFF within the time frame of the study when randomized in the control group
* Finally, the participating hospitals need an expected volume of more than one hundred COPD-exacerbation or PFF patients annually.
* To have a comparable sample across all clusters, the following inclusion criteria on individual level are set:

  1. All professionals that according to the medical head of the division and head nurse are member of the interprofessional team caring for COPD-exacerbation or PFF patients from admission until discharge out of the acute hospital ward
  2. To be part of the interprofessional care team is further conceptualized as being part of the group of clinicians and staff who have a shared clinical purpose and direct care responsibilities for the respective patient group during the set time period
  3. All individual participants need to be member of the team during one specific week, where patients are being followed for the two other trials of the EQCP-project (8). This specific week is chosen by the study coordinator and can be defined as an average week, with normal staff ratios
  4. Because we want to study interprofessional teamwork, each cluster is asked to minimally include the orthopedic surgeons/pneumologists, head nurse, nurses, physiotherapists and social workers in their sample. Based on their own judgment, the chief medical doctor, in consensus with the head nurse, can decide to include other professional groups in their sample
  5. In some hospitals COPD-exacerbation or PFF patients are being admitted at multiple nursing wards, e.g. due to capacity problems or other organizational issues. If that is the case, then the clusters are asked to only include these team members that are working on the ward where the respective patient groups are being admitted most frequently.

Exclusion Criteria:

* All team members that are not working (e.g. on leave) during the chosen week
* All team members who are only temporarily part of the team (e.g. student nurses in training).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2009-05; Primary Completion 2014-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Relational Coordination | For average period of 3 months
  Relational coordination describes the quality of communication and functional relations within a interprofessional team with shared goals and interdependent tasks.

SECONDARY OUTCOMES:
Perceived Organisation of Care | For average period of 3 months
  The perceived organisation of care is a team indicator to measure the actual organisation of the care process. It is measured in a valid and reliable way by using the Care Process Self Evaluation Tool (CPSET).
Work engagement | For average period of 3 months
  Work engagement is a measure to analyse the level of competence, emotional exhaustion and mental detachement measured with the Burnout Inventory.
Team Climate | For average period of 3 months
  Team climate is an indicator to measure the team vision, participative safety, support for innovation and task orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, PhD, Study Director — KU Leuven; Walter Sermeus, PhD, Principal Investigator — KU Leuven; Massimiliano Panella, PhD, Principal Investigator — Amedeo Avogadro University of Eastern Piemont; Svin Deneckere, MSc, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Deneckere S, Robyns N, Vanhaecht K, Euwema M, Panella M, Lodewijckx C, Leigheb F, Sermeus W; EQCP-studygroup. Indicators for follow-up of multidisciplinary teamwork in care processes: results of an international expert panel. Eval Health Prof. 2011 Sep;34(3):258-77. doi: 10.1177/0163278710393736. Epub 2010 Dec 29. PMID 21190951
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Deneckere S, Euwema M, Lodewijckx C, Panella M, Sermeus W, Vanhaecht K. The European quality of care pathways (EQCP) study on the impact of care pathways on interprofessional teamwork in an acute hospital setting: study protocol: for a cluster randomised controlled trial and evaluation of implementation processes. Implement Sci. 2012 May 18;7:47. doi: 10.1186/1748-5908-7-47. PMID 22607698
- See also: European Pathway Association — http://www.E-P-A.org